CLINICAL TRIAL: NCT00140647
Title: The Study of Atherosclerosis With Ramipril and Rosiglitazone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gerstein, Hertzel, MD (Individual)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: STARR
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Atherosclerosis; Impaired Glucose Tolerance; Isolated Impaired Fasting Glucose; Cardiovascular Disease
Keywords: atherosclerosis; carotid artery; ramipril; rosiglitazone; impaired glucose tolerance; impaired fasting glucose; diabetes prevention
MeSH Terms: conditions — Atherosclerosis; Glucose Intolerance; Cardiovascular Diseases | interventions — Ramipril; Rosiglitazone

INTERVENTIONS:
Drug: Ramipril
Drug: Rosiglitazone

SUMMARY:
The purpose of this study is to determine if ramipril and/or rosiglitazone retard the progression of atherosclerosis as evaluated by serial carotid intermedial thickness measurements.

DETAILED DESCRIPTION:
STARR is a multi-centre, international, randomized controlled clinical trial with a 2x2 factorial design, that will evaluate the effects of ramipril and of rosiglitazone on atherosclerosis progression, as determined by B-mode carotid ultrasound (US). It is designed as a substudy of DREAM (Diabetes Reduction Assessment with ramipril and rosiglitazone Medications) Trial. The study is designed to enroll 1,200 study participants and follow is proposed for an average of 3.75 years.

SIGNIFICANCE OF THE PROPOSED RESEARCH: With regards to ramipril this study will provide important mechanistic data regarding potential benefits of ACE inhibitor therapy on atherosclerosis and by inference in reducing CV risk in a lower risk younger population than studied in previous trials. In this population a clinical outcome trial focusing primarily on CV events would be difficult to conduct due to the expected fairly low event rate. If the study on atherosclerosis is positive, this may provide a rational for therapy in this subset of patients without overt CVD or diabetes, but with impaired glucose tolerance or impaired fasting glucose.

ELIGIBILITY:
Inclusion Criteria:

* impaired glucose tolerance (FPG < 7 mmol/L or 126 mg/dL & 2hr PG between 7.8-11.0 mmol/l [140-199 mg/dl] after a 75 g OGTT
* impaired glucose tolerance (FPG≥ 6.1 mmol/l [110 mg/dl]) and no diabetes (i.e. a FPG < 7.0 mmol/l [126 mg/dl])
* a technically adequate baseline carotid ultrasound examination

Exclusion Criteria:

* current use of an ACE-inhibitor (ACE-I) or thiazolidinedione (TZD)
* known hypersensitivity to ACE-I
* prior use of anti-diabetic medications 9with the exception of during pregnancy)
* use of systemic glucocorticoids or niacin
* congestive heart failure or EF < 40%
* existing cardiovascular disease (previous MI, stroke, angina, uncontrolled hypertension)
* diabetes
* renal or hepatic disease
* major illness
* use of another experimental drug
* pregnant or unwilling to use reliable contraception
* major psychiatric disorder
* diseases that affect glucose tolerance
* unwillingness to be randomized or sign informed consent
* known uncontrolled substance abuse
* inability to communicate with research staff

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200
Dates: Start 2001-07; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
The change of the mean maximum carotid intimal medial thickness (IMT)evaluated across 12 segments involving the left and right common carotid, bifurcation and internal carotid arteries.

SECONDARY OUTCOMES:
The change over time in the mean IMT across the common carotid far wall IMT of the right and the left carotid arteries.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Lonn, MD, Principal Investigator — McMaster University

REFERENCES:
- [Derived] Lonn EM, Gerstein HC, Sheridan P, Smith S, Diaz R, Mohan V, Bosch J, Yusuf S, Dagenais GR; DREAM (Diabetes REduction Assessment with ramipril and rosiglitazone Medication) and STARR Investigators. Effect of ramipril and of rosiglitazone on carotid intima-media thickness in people with impaired glucose tolerance or impaired fasting glucose: STARR (STudy of Atherosclerosis with Ramipril and Rosiglitazone). J Am Coll Cardiol. 2009 Jun 2;53(22):2028-35. doi: 10.1016/j.jacc.2008.12.072. PMID 19477351